CLINICAL TRIAL: NCT01818310
Title: Randomised Clinical Study of Safety and Efficacy of Autologous Bone Marrow Aspirate Concentrate (BMAC) for No-option_critical Limb Ischemia in Type-II Diabetes Mellitus Patients. (DIALEG)
Brief Title: Safety and Efficacy Study of Autologous Bone Marrow Aspirate Concentrate for No-Option Critical Limb Ischemia
Acronym: DIALEG
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government); Regional Council of the Moravian-Silesian region, KU MSK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-T2DM-CLI; 2012-001825-28 (EudraCT Number)
Record Dates: First submitted 2012-09-27; First posted 2013-03-26 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Critical Lower Limb Ischemia; Type-2 Diabetes Mellitus
Keywords: ischemia; diabetes mellitus; bone marrow aspirate concentrate (BMAC)
MeSH Terms: conditions — Ischemia; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A: Intramuscular (Experimental): Intramuscular BMAC application The study subjects in the Group A will receive a treatment of 35ml BMAC administered intramuscularly into the affected limb, in individual punctures of 1 ml.
  The punctures will be applied into the crural muscle around the defect, the procedure takes approx. 60 minutes.
  Interventions: Biological: Group A: Intramuscular
- Group B: Intraarterial (Experimental): Intraarterial BMAC application The study subjects in the Group B will receive a treatment of 35ml BMAC administered intraarterially into the affected limb.
  Interventions: Biological: Group B: Intraarterial
- Group C: Intravenous (Experimental): Group C: Intravenous The study subjects in the Group C will receive a treatment of 35ml BMAC administered intravenously into the affected limb.
  Interventions: Biological: Group C: Intravenous
- Group D: Control-standard treatment (Other): Group D: Control Group Study subjects in Group D will receive a standard treatment for NO-option CLI.
  Interventions: Procedure: Group D: Surgical endovascular treatment with maximum medicamentous treatment

INTERVENTIONS:
Biological: Group A: Intramuscular — Intramuscular BMAC application The study subjects in the Group A will receive a treatment of 35ml BMAC administered intramuscularly into the affected limb, in individual punctures of 1 ml.
  The punctures will be applied into the crural muscle around the defect, the procedure takes approx. 60 minutes.
  Arms: Group A: Intramuscular
Biological: Group B: Intraarterial — Intraarterial BMAC application The study subjects in the Group B will receive a treatment of 35ml BMAC administered intraarterially into the affected limb.
  Arms: Group B: Intraarterial
Biological: Group C: Intravenous — Group C: Intravenous The study subjects in the Group C will receive a treatment of 35ml BMAC administered intravenously into the affected limb.
  Arms: Group C: Intravenous
Procedure: Group D: Surgical endovascular treatment with maximum medicamentous treatment — Group D: Control Group Control Group - no experimental intervention, standard endovascular treatment or bypass surgery or maximum medicamentous treatment
  Arms: Group D: Control-standard treatment

SUMMARY:
The aim of the presented clinical trial is to evaluate a hypothesis, that BMAC prepared from bone marrow aspirate and injected intramuscularly into ischemic areas of the lower extremity in patients with diabetes mellitus type II., intraarterially into the defect of the limb or with an intravenous application only, has a greater potential to improve the perfusion in the ischemic limbs than standard treatment of NO-CLI. Another aim of the study is to find out differences among three different therapeutic types of BMAC application, to define their effectiveness and safety and to compare the impact of different means of application to the speed of healing of the limb defects and the improvement of perfusion parameters.

DETAILED DESCRIPTION:
Secondary hypothesis assumes, that the intravenous application of BMAC in patients with T2DM older than 30 years of age, with a dose of insulin exceeding 0.7 U/kg/day or 50U/day will result in decreasing the insulin dose in the course of 6-month follow-up and in an improvement of the glycHBA1c levels, improvement of the liver and kidney function, decrease of the cholesterol levels and improvement of the immune response parameters, i.e. parameters of lymphocytar blastic transformation, more than in case of patients with intramuscular or intraarterial application of BMAC.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* diagnosis of critical limb ischemia
* non-healing defect on the study limb
* ABI value < 50 mmHg or ABI< 0.4
* TBI value < 40 mmHg or TBI < 0.4
* TcPO2 < 20 mmHg in supine position
* no other suitable surgical or re-vascularization procedure
* age > 18 years
* signed Informed Consent

Exclusion Criteria:

* non-signing of the Informed Consent
* anticipated life expectancy < 6 months
* history of bone-marrow disease
* renal failure or dialysis dependency
* known malignant disease
* health risks excluding the possibility of general anaesthesia or sedation
* life-threatening ischaemic heart disease
* vast necrosis of the index limb
* active infectious disease, or ATB treatment
* treatment with immunosupressives
* pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Amputation-free survival | 18 months
  The data for Primary outcome will be collected throughout the first 18 months of the study. The assessed parameters will include amputation-free survival in order to verify the safety and efficacy of the treatment.

SECONDARY OUTCOMES:
Tissue perfusion parameters | 4 years
  The efficacy of BMAC application will be evaluated throughout the whole course of the clinical trial, with final assessment at the end of the trial.
  * Increase of the monitored parameters of the tissue perfusion measured with LDP-Periflux 5000 (Perimed), i.e. increase of the ABI - ankle-brachial index, TP - toe pressure, TBI- Toe Brachial index and TcpO2- transcutaneous oxygen pressure.
  * Decrease of the SPP perfusion parameter - skin perfusion pressure reflecting an inflammatory activity of the affected limb.
Clinical outcome classification | 4 years
  The efficacy of BMAC application will be evaluated throughout the whole course of the clinical trial, with final assessment at the end of the trial.
  - Improvement of the Rutherford scale of CLI
Functional angiogenesis imaging outcome | 4 years
  The efficacy of BMAC application will be evaluated throughout the whole course of the clinical trial, with final assessment at the end of the trial.
  - Increase of the number and quality of newly created vessels measured according to digital subtraction angiography (DSA) or MR-angiography (in allergic patients)
Quality of life outcome | 4 years
  The efficacy of BMAC application will be evaluated throughout the whole course of the clinical trial, with final assessment at the end of the trial.
  * Measurable decrease of pain measured on the scale and QOL questionnaire (RAND-36).
  * Healing of the defect or gangrene (size and state of the wound)

OTHER OUTCOMES:
Changes in lymphocyte subsets and levels of inflammatory and antiinflammatory cytokines in each of the groups. | 24 months
  The immune response of study subjects will be monitored following the transplantation of stem cells, together with the periphery lymphocyte function (T-cells, B-cells, NK-cells).
  Immune response parameters, (i.e. parameters of lymphocytar blastic transformation)
Metabolic response | 24 months
  The following laboratory parameters throughout the clinical trial:
  * liver and kidney function
  * lipid spectra
Blood glucose and pancreatic function response | 24 months
  The following parameters will be monitored in the study subjects:
  * glycHBA1c levels
  * C-peptide

CONTACTS AND LOCATIONS:
Overall Officials: Vaclav Prochazka, MD, PhD, MSc, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dormandy J, Heeck L, Vig S. The natural history of claudication: risk to life and limb. Semin Vasc Surg. 1999 Jun;12(2):123-37. PMID 10777239
- [Background] Clair DG, Dayal R, Faries PL, Bernheim J, Nowygrod R, Lantis JC 2nd, Beavers FP, Kent KC. Tibial angioplasty as an alternative strategy in patients with limb-threatening ischemia. Ann Vasc Surg. 2005 Jan;19(1):63-8. doi: 10.1007/s10016-004-0136-0. PMID 15714369